CLINICAL TRIAL: NCT02602418
Title: Neural Correlates of Working Memory Training for HIV Patients: A Randomized Control Clinical Trial
Brief Title: Neural Correlates of Working Memory Training for HIV Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Hawaii (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Linda Chang, M.D., Professor, University of Maryland, College Park
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4R01DA035659-04 (NIH); 4R01DA035659-04 (NIH)
Record Dates: First submitted 2015-11-05; First posted 2015-11-11 (Estimated); Last update posted 2019-10-02 (Actual); Status verified 2019-10

CONDITIONS: HIV Infection
Keywords: Human Immunodeficiency Virus (HIV); working memory training; brain function; functional magnetic resonance imaging (fMRI)
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HIV Positive participants (Experimental): Intervention; 90 HIV positive participants will be trained. Half the participants will have the Adaptive WM Cogmed training, and half will have the non-adaptive WM Cogmed training.
  Interventions: Other: Adaptive WM CogMed Training; Other: Nonadaptive WM CogMed Training
- Seronegative particpiants (Other): Intervention; 90 seronegative participants will be trained. Half the participants will have the Adaptive WM Cogmed training, and half will have the non-adaptive WM Cogmed training.
  Interventions: Other: Adaptive WM CogMed Training; Other: Nonadaptive WM CogMed Training

INTERVENTIONS:
Other: Adaptive WM CogMed Training — 12 different computerized visual and spatial Working Memory tasks will be presented at each sessoin. Each session will involve 8 of the 12 tasks, and each subject is required to complete 25 training sessions, 30-40 minutes per day, 4-5 days per week over a 5-8 week period (minimum 20 sessions). The tasks will become more difficult in an "adaptive" manner, which is hypothesized as optimal for learning and training effects.
Other: Nonadaptive WM CogMed Training — The same 12 computerized visual and spatial working memory tasks will be presented, but at a fixed ("non-adaptive") and low difficulty level. 5 sessions per week x 5 weeks fora total of 25 sessions (minimum 20 sessions).

SUMMARY:
Despite potent combination antiretroviral therapy, cognitive (memory and concentration) problems continue to occur in up to 50% of HIV-infected individuals, especially in older infected individuals, and those who abuse alcohol, marijuana or psychostimulants. Since no effective treatments are available to these individuals with cognitive problems, conservative estimates indicate that the cost of care for these patients could double in the next two decades. To address this urgent problem, this study will use a comprehensive approach (cognitive tests, functional MRI and several biomarkers) to evaluate whether a novel computer-based training program would improve the brain function, especially working memory and attention, in HIV-infected and infected individuals.

DETAILED DESCRIPTION:
The Overall Goals are to perform a double blind placebo-controlled study using Cogmed™ to determine whether this adaptive WM training program will benefit HIV-infected individuals, and whether the investigators can identify individuals who might benefit most from the working memory (WM) training. Lastly, the investigators will explore how brain activation, neuroinflammation and cerebrospinal fluid (CSF) monoamine levels might be related to WM function before and after the training.

ELIGIBILITY:
Inclusion Criteria for HIV-infected participants :

1. Men or women of any ethnicity, ages>18 years and able to provide informed consent,
2. HIV seropositive (with documentation from medical records),
3. Stable on an antiretroviral regimen for 6 months or will remain without antiretroviral treatment during the duration of the study.

Inclusion Criteria for Seronegative (SN) healthy participants :

1. Men or women of any ethnicity, ages > 18 years and able to give informed consent,
2. Seronegative for HIV

Exclusion criteria :

1. Confounding co-morbid psychiatric illness
2. Confounding neurological disorders
3. Abnormal screening laboratory tests (>2 SD) that might indicate a chronic medical condition (e.g. diabetes, severe cardiac, renal or liver disorders)
4. Medications that might influence outcome measures
5. Current or history of drug dependence within the past two years
6. Positive urine toxicology screen
7. Inability to read at an 8th grade level
8. Other contraindications for MR studies

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2012-09 (Actual); Primary Completion 2020-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Changes in the Improvement Index on Cogmed™ | 1 month after training, and 6 month after training completion
  This is generated by the computer training program based on the trained tasks.
Changes in Performances on near transfer working memory tasks | 1 month after training, and 6 month after training completion
  Verbal working memory and spatial working memory tasks
Changes in Blood-Oxygenation Level-Dependent Functional MRI Measures | 1 month after training, and 6 month after training completion
  Brain activation during the performance of working memory and attention tasks

SECONDARY OUTCOMES:
Changes in cognitive performance based on LIM homeobox transcription factor 1 alpha (LMX1A) genotypes (AA vs. GA/GG) | Baseline, 1 month after training, and 6 month after training completion
  Performance and improvements on cognitive tests may vary at baseline and after training based on LMX1A genotypes
Changes in Behavior Rating Inventory of Executive Function-Adult Version (BRIEF-A) | 1 month after training, and 6 month after training completion
  Improvement on BRIEF-A, a self-reported evaluation of the person's executive function during their activities of daily living.
Changes in Blood-Oxygenation Level-Dependent Functional MRI Measures based on LMX1A genotypes | 1 month after training, and 6 month after training completion
  Brain activation during working memory performance may vary at baseline, 1-month or 6-months based on the different LMX1A genotypes

CONTACTS AND LOCATIONS:
Overall Officials: Linda Chang, MD, Principal Investigator — University of Maryland Baltimiore
Locations (1):
- University of Maryland School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chang L, Liang H, Ernst T, Cunningham E, Wang J, Baptiste J, Lohaugen GCC. LMX1A and APOE varepsilon Genotype Associations With Working Memory Training Effects in HIV and Non-HIV: A Randomized Controlled Trial. Neurol Neuroimmunol Neuroinflamm. 2026 Jan;13(1):e200519. doi: 10.1212/NXI.0000000000200519. Epub 2025 Dec 11. PMID 41380114
- [Derived] Chang L, Lohaugen GC, Douet V, Miller EN, Skranes J, Ernst T. Neural correlates of working memory training in HIV patients: study protocol for a randomized controlled trial. Trials. 2016 Feb 2;17:62. doi: 10.1186/s13063-016-1160-4. PMID 26833223